CLINICAL TRIAL: NCT00472394
Title: Determining Women's Preferences for Medical Abortion Using Willingness to Pay
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Other Study IDs: WTP
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Medical Abortion
Keywords: Medical abortion; Preferences; Willingness to Pay

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
New medical abortion regimens are being tested with increasing frequency. However women's preferences for certain attributes of the regimes are not being investigated to any great degree. Consideration of women's preferences in designing new regimens may help to optimize the medical abortion process. The proposed prospective survey research will attempt to determine women's preferences for individual aspects of medical abortion treatment and various regimens, and to determine what attributes of medical abortion treatment may be driving these preferences. The information collected in this study may be used in developing future treatment regimens or as the groundwork for future research into preferences, acceptability, and satisfaction with treatment.

DETAILED DESCRIPTION:
The FDA-approved regimen for medical abortion specifies treatment with oral mifepristone followed 48 hours later by oral misoprostol. Women's experiences with this regimen were assessed in the early medical abortion trials that preceded FDA approval. The majority of women who used this regimen rated their experience as satisfactory or very satisfactory after the abortion was completed (Newhall 2000). A weakness of these data is that they were collected from women who likely had an a priori preference for medical abortion as demonstrated by their participation in experimental studies of this method. Other factors affecting women's preferences had little to do with medical abortion per se such as the ability to avoid the involvement of their insurance company by participating in a study or that the method was offered free of charge (Clark S, et al. 2000).

Since the time that these studies were performed, multiple investigations have evaluated alternative regimens of using mifepristone and misoprostol for medical abortion (Creinin MD, 2000). Improving efficacy, reducing side effects, and increasing the flexibility in the timing and route of medication administration have driven the development of these alternative regimens (Newhall EP and Winikoff B, 2000).

As with earlier studies, most trials of new regimens have assessed acceptability or satisfaction post-treatment. In general, overall satisfaction has been reported as high regardless of regimen (Ho PC, 2006). However, when asked about specific aspects of the medical abortion treatment, women's preferences appear to be more nuanced. Route of misoprostol administration is one example. Shannon, et al. (2006) compared mifepristone with oral or vaginal misoprostol and found an overall acceptability of 91%, regardless of route of administration. However, when specifically asked about preference for route, the odds of preferring oral administration greatly exceeded the odds of preferring vaginal (OR = 13.7, 95% CI 6.5-28.7). A preference for oral administration was also demonstrated in a comparative trial by Schaff, et al. (2001), however this preference was driven by the greater amount of pain experienced by the vaginal group.

Further insight into the complexity of acceptability and satisfaction with specific regimens was provided by a pilot study that I performed of mifepristone and buccal misoprostol (4 tablets of misoprostol dissolved between the cheek and gum for 30 minutes). Detailed information regarding acceptability, likes, and dislikes was collected pre- and post-treatment. As with other studies, 91% of women surveyed would choose medical abortion again. However, only 42% found the experience to be a positive one. When asked specifically about the buccal route of administration, 72% disliked some aspect of using misoprostol in this way. Of note, pre-treatment, just under half of the women would have preferred oral administration and 13% buccal. Post-treatment, women were asked which route they would prefer assuming equal efficacy. The majority (70%) listed oral whereas the preference for buccal dropped to 9%. Most women cited dissatisfaction with the experience of using misoprostol buccally either because it was inconvenient, tasted bad, or had a chalky aftertaste.

Questions about preferences usually include an assumption that all factors other than the specific attribute being examined are equal, which may or may not be the case. Careful examination of specific regimens presented as part of comprehensive scenarios joined with use of targeted questions may provide more insight into our lack of understanding of preferences. It is still unclear, for example, what decrement in efficacy, and subsequent need for a surgical procedure, in combination with what degree of expected side effect and expected amount of pain, and which route and timing of administration, women would find acceptable and thus would determine their preferences if all of the options were available to them.

The purpose of this study is to ascertain women's preferences for different aspects of medical abortion treatment. In addition to questions directly assessing preferences, the economic instrument of willingness to pay (WTP) will be employed. The technique of WTP is based on the premise that the maximum amount of money an individual is willing to pay for an attribute of treatment is an indicator of the utility or satisfaction to her of that attribute (Donaldson C, 1993). This method has been used successfully in measuring the strength of preference for medical or surgical abortion (Gibb S, et al. 1998), miscarriage management (Ryan and Hughes, 1997), and models of antenatal care (Ryan M, et al., 1997). As opposed to "strength of preference" measures that use a scale of quality adjusted life years, which involve a time trade-off to achieve an improvement in a state of being, WTP values health options by placing a monetary value on each option (Gibb, 1998). The maximum WTP can be taken as an indication of preference strength for one option over another and relative WTP values can be meaningfully compared assuming a like unit of measurement, for example of oral versus vaginal misoprostol administration.

The proposed survey addresses the characteristics of the FDA approved-regimen and alternative regimens that have been designed and studied thus far. The variables included are the mode of misoprostol administration (oral, buccal, vaginal, and sublingual), the time lapse between mifepristone and misoprostol administration, where the medications will be taken (at home compared with in the physician's office), side effects, pain, and efficacy. We have attempted to be as inclusive as possible regarding the modifiable attributes of medical abortion treatment such as route or timing of medication administration. The survey is divided into three sections. The first section utilizes the WTP methodology in scenarios about side effects and comparisons of different medical abortion regimens, and includes a single overall comparison of medical with surgical abortion. With regard to the medical regimens, the FDA-approved regimen, buccal, sublingual, and oral alternative regimens are all compared with the vaginal regimen that is most commonly used in the United States today. The values used in each regimen's side effect, pain, and efficacy profiles are based on gestational age appropriate results from clinical trials. For example, the FDA-approved regimen is only for use through seven weeks of gestation. It was, therefore, compared with the vaginal regimen as it performs through seven weeks. Similarly, the buccal alternative has only been studied in a randomized controlled trial against the vaginal regimen though eight weeks of gestation.

The second section of the survey asks women to rank and rate individual characteristics of medical abortion treatment that are presented in the scenarios. The ranking and rating questions serve two purposes, 1) convergent validity can be determined when comparing the dollar amounts given in the WTP questions (implicit ranking) compared with the explicit rankings and ratings given in the other questions and 2) they address individual variables that are encompassed within each WTP scenario in an attempt to tease out how preferences for certain aspects of medical abortion regimens compare to each other and which aspects might be determining preferences.

The third section collects demographic data, including income level, as well as pregnancy and previous abortion history.

New medical abortion regimens are being tested with increasing frequency; however women's experiences with these regimens are not being explored to any great degree. Consideration of women's preferences in designing new regimens may help optimize the medical abortion process. This prospective evaluation will attempt to determine which aspects of medical abortion treatment women value, and thus prefer, most. The information collected in this study may be used as a guide in developing future treatment regimens or clinical protocols.

Design and methodology

Women, 18 years of age or older, who present to the Center for Family Planning Research (CFPR) at Magee-Womens Hospital desiring a medical abortion will be invited to participate in this study. The anticipated sample size is approximately 200. The attached survey (see Attachment 1) will be given to each subject willing to participate in the study prior to any screening procedures for her abortion. All subjects will be introduced to the survey content, intent, and methods in a face-to-face discussion with a research assistant. The subjects will then be given time to complete the survey independently. Research assistants will be available for technical guidance or to answer technical questions as needed. Subjects will complete this one-time survey anonymously. After the survey is completed the subjects will be screened and the abortion performed.

Data analysis

Collected data from the questionnaires will be compiled and descriptive statistics will be generated. Maximum willingness to pay (WTP) values will be estimated using the mean and median. Association and difference comparisons of categorical values will be made using Chi-square and Fisher's exact test where appropriate and continuous values using Student's t-test. Univariable and multivariable regression analysis will be performed to determine predictors of preferences based on WTP.

Finally, preference and demographic data will be used to create a regression model to evaluate what, if any, discrete factors drive women's preferences. This model also will be used to adjust WTP values so that they can be taken as indications of willingness to pay and not ability to pay.

Number of subjects and statistical power

The study population will be a non-probability based convenience sample of women presenting to the CFPR for medical abortion from October, 2006-April, 2007. It is estimate that approximately 200 women will be able to complete the survey during this time. The number is estimated based on our currently ongoing medical abortion trial, which will include 175 women, as well as those women undergoing non-trial related medical abortions through our office. All women presenting to the Center for a medical abortion will be informed of the survey and it is anticipated that most will be willing to participate. It is unclear what proportion of subjects will prefer which medical abortion attributes. Using a conservative proportional estimate of .5, a probability sample size of 200 gives a 90% confidence level with a margin of error of 6%.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged 18 years or older, who present to the Center for Family Planning Research desiring a medical abortion and are able to read English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2006-10; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Lohr, MD, Principal Investigator — University of Pittsuburgh
Locations (1):
- Center for Family Planning Research, Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States